CLINICAL TRIAL: NCT04937894
Title: The Efficacy and Safety of Tigecycline for the Treatment of Infectious Diseases
Brief Title: Antibiotic Therapy for Infectious Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Collaborators: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Wei Zhao, Head of department of clinical pharmacy and pharmacology, Shandong University
Other Study IDs: 2021_TIG_001
Record Dates: First submitted 2021-06-17; First posted 2021-06-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Infectious Disease
MeSH Terms: conditions — Communicable Diseases | interventions — Tigecycline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Tigecycline — Efficacy and safety of Tigecycline

SUMMARY:
Tigecycline is a last-resort antibiotic that is used to treat severe infections caused by extensively drug-resistant bacteria. However, the efficacy and safety data for tigecycline in infectious patients are lacking. The aim of this study is to assess the efficacy and safety of tigecycline in infectious patients using pharmacokinetics and omics.

ELIGIBILITY:
Inclusion Criteria:

* critically ill hospitalized males or nonpregnant females aged 18 years with severe infections which the treating clinician was treating with tigecycline

Exclusion Criteria:

1. severe liver dis- eases (e.g., Child-Pugh score C);
2. patients allergic to tetracycline and tigecycline;
3. those who have participated in other clinical trials, or those who are considered unsuitable by researchers;
4. pregnant women and lactating women.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with severe infections
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Through study completion, an average of 15 days
  Drug-related adverse events and serious adverse events
Pharmacokinetics of tigecycline | Through study completion, an average of 3 days
  clearance in L/h
Rate constant for tigecycline distribution | Through study completion, an average of 3 days
  Pharmacokinetics of tigecycline
The ratio of area under the concentration-time curve (AUC) to minimum inhibitory concentration (MIC). | Through study completion, an average of 3 days
  PD target

SECONDARY OUTCOMES:
fibrinogen levels in mg/dL | Through study completion, an average of 3 days
prothrombin time | Through study completion, an average of 3 days
  prothrombin time in second
activated partial thromboplastin time | Through study completion, an average of 3 days
  activated partial thromboplastin time in second
international normalized ratio | Through study completion, an average of 3 days
  international normalized ratio，INR
blood platelet count | Through study completion, an average of 3 days
  blood platelet count in ×10^9/L
thrombin time | Through study completion, an average of 3 days
  thrombin time in second

CONTACTS AND LOCATIONS:
Locations (1):
- Wei Zhao, Jinan, Shandong, China